CLINICAL TRIAL: NCT06032559
Title: Implementation and Effectiveness of Mindfulness Oriented Recovery Enhancement as an Adjunct to Methadone Treatment for Opioid Use Disorder and Chronic Pain
Brief Title: Implementation and Effectiveness of Mindfulness Oriented Recovery Enhancement as an Adjunct to Methadone Treatment
Acronym: IMPOWR-MORE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Utah (Other)
Responsible Party: Principal Investigator, Nina A. Cooperman, Psy. D., Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro2022001626; R01DA056537 (NIH)
Record Dates: First submitted 2023-09-04; First posted 2023-09-13 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Opioid Use; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- MORE (Experimental): Eight group sessions of Mindfulness-Oriented Recovery Enhancement plus methadone treatment as usual (TAU)
  Interventions: Behavioral: MORE
- Scripted Mindfulness Practice (SMP) (Active Comparator): Eight group sessions of scripted mindfulness practice plus TAU.
  Interventions: Behavioral: SMP
- Treatment-as-Usual (Active Comparator): Methadone treatment as usual.
  Interventions: Other: TAU

INTERVENTIONS:
Behavioral: MORE — MORE plus TAU
  Arms: MORE
Behavioral: SMP — SMP plus TAU
  Arms: Scripted Mindfulness Practice (SMP)
Other: TAU — TAU only
  Arms: Treatment-as-Usual

SUMMARY:
This hybrid implementation-effectiveness trial will evaluate Mindfulness-Oriented Recovery Enhancement (MORE) for patients with opioid use disorder receiving methadone treatment (MT). The investigators will also assess barriers and facilitators to integrating MORE into methadone treatment, and evaluate the impact of a sustainable train-the-trainer model on provider burden, intervention fidelity, intervention engagement, and outcomes. Participants will be assigned to a higher intensity MORE implementation strategy, a minimal intensity implementation strategy consisting of a simple, scripted mindfulness practice (SMP) extracted from the MORE treatment manual with minimal training and feedback and no supervision, or methadone treatment as usual (TAU). We aim to:

* Examine barriers and facilitators to the implementation of MORE and SMP in MT and evaluate strategies for optimizing training, fidelity, and engagement.
* Evaluate the effectiveness and treatment fidelity of a higher intensity MORE implementation strategy versus a lower intensity, scripted mindfulness practice (SMP) implementation strategy as an adjunct to methadone TAU or methadone TAU, only. Outcomes include opioid and other drug use, craving, MT discontinuation, depression, anxiety, and physical pain (secondary outcomes) than patients randomized to TAU.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* age ≥18
* currently on methadone
* persistent or recurring pain that has lasted for a duration of 3 months of longer.

Exclusion Criteria:

* severe cognitive impairment (score >23 on Mini Mental Status Exam) or psychosis (positive SCID Psychotic Screen)
* suicidal risk (score ≥7 on Suicidal Behaviors Questionnaire)
* inability to attend or fully participate in intervention sessions or assessments
* previous formal mindfulness training (e.g., MBSR, MBRP) or MORE (from the R21 or R33 studies).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Days of drug use | Baseline through 52 weeks
  mber of days of drug use as measured by self-reported days of use and biochemically verified use via drug screen.

SECONDARY OUTCOMES:
Chronic Pain | Baseline through 52 weeks
  Chronic pain measured by the Brief Pain Inventory Short Form (range 0-10, with higher scores indicating worse pain).

CONTACTS AND LOCATIONS:
Overall Officials: Eric Garland, Ph, Principal Investigator — Rutgers Robert Wood Johnson Medical School
Locations (2):
- United States (2):
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
All participant data collected during the trial will be shared after de-identification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 3 months and ending five years after study publication.
Access Criteria: Researchers who provide a methodologically sound proposal.